CLINICAL TRIAL: NCT05069779
Title: The Acute Effects of Diazepam on Blood Pressure Regulation
Brief Title: Diazepam and Blood Pressure Regulation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 70101717.1.0000.5103
Record Dates: First submitted 2021-09-15; First posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Healthy
Keywords: Blood pressure; Benzodiazepine; Autonomic nervous system
MeSH Terms: interventions — Diazepam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Diazepam (Experimental): Oral
  Interventions: Drug: Diazepam
- Placebo (Placebo Comparator): Oral
  Interventions: Drug: Diazepam

INTERVENTIONS:
Drug: Diazepam — Oral administration of 10 mg of diazepam

SUMMARY:
The aim of this study is to determine the acute effects of diazepam on beat-to-beat blood pressure variability and baroreflex control.

DETAILED DESCRIPTION:
Benzodiazepines are widely prescribed for a variety of clinical conditions. However, its cardiovascular consequences remain controversial. In this study, the investigators sought to determine the acute effects of a single dose of oral diazepam (10mg) on resting beat-to-beat blood pressure variability and cardiac and sympathetic baroreflex sensitivity in a cohort of young, healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 40 years of age
* Healthy, free of known cardiovascular, metabolic, or musculoskeletal disease

Exclusion Criteria:

* History of smoking (tobacco or cannabis), defined as any smoking within the past 3 months
* Diagnosed cardiovascular or metabolic disease(s)
* Prescription of chronic medications other than oral contraceptives
* History of hypertension or presence of arrhythmia

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Resting beat-to-beat blood pressure variability | Change from baseline at 60 min
  Finger photoplethysmography
Systolic and diastolic blood pressure | Change from baseline at 60 min
  Oscillometric device

SECONDARY OUTCOMES:
Muscle sympathetic nerve activity | Change from baseline at 60 min
  Microneurography
Baroreflex sensitivity | Change from baseline at 60 min
  The relationship between changes in beat-to-beat blood pressure and heart rate (cardiac baroreflex) or MSNA (sympathetic baroreflex).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Brasilia, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The data underlying this project will be shared on reasonable request to the principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR